CLINICAL TRIAL: NCT03328299
Title: Pharmacokinetics and Dynamics of Dexmedetomidine as Adjuvant in TAP Block for Patient Undergoing Lower Abdominal Surgery
Brief Title: Pharmacokinetics and Dynamics of Dexmedetomidine as Adjuvant in TAP Block
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Adel El sherif,MD, lecturer of anesthesia , ICU and pain management, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 402
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine group (Active Comparator): patients were given ultrasound guided TAP-block with 20 ml of 0.5 % bupivacaine + dexmedetomidine 1 μg•kg-1 diluted in 20 ml saline
  Interventions: Drug: Dexmedetomidine
- bupivacaine group (Placebo Comparator): patients will given ultrasound guided TAP-block with 20 ml of 0.5 % bupivacaine
  Interventions: Drug: bupivacaine

INTERVENTIONS:
Drug: Dexmedetomidine — 20 ml of 0.5 % bupivacaine plus dexmedetomidine 1 μg•kg-1
  Other Names: active group
  Arms: Dexmedetomidine group
Drug: bupivacaine — 20 ml of 0.5 % bupivacaine
  Other Names: control
  Arms: bupivacaine group

SUMMARY:
TAP-block has been shown to be a safe and effective postoperative analgesia method in a variety of general. Dexmedetomidine is a selective α2 agonist with 8 times more affinity for α2 adrenergic receptors compared to clonidine and possesses all the properties of α2 agonist without respiratory depression. Dexmedetomidine has been focus of interest for its broad spectrum (sedative, analgesic and anesthetic sparing) properties, making it a useful and safe adjunct in many clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* 24 ASA I-II
* patients (age 18-60 years
* weight 50-89 kg

Exclusion Criteria:

* a known allergy to the study drugs
* significant cardiac
* respiratory, renal or hepatic diseases
* bleeding diathesis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2017-11-11 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
measure dexmedetomidine level into systemic circulation after local administration | up to 6 hours
  assessment of systemic dexmedetomidine level after local administration in TAP block after 15 minutes after giving the block, 30 min, 45 min, 1hrs, 2hrs, 4hrs and 6

SECONDARY OUTCOMES:
total dose of IV PCA morphine consumption in the first 24 h postoperative | 24 hours
  postoperative morphine consumption

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer instIitute, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El Sherif FA, Abdel-Ghaffar H, Othman A, Mohamed S, Omran M, Shouman S, Hassan N, Allam A, Hassan S. Pharmacokinetics and Pharmacodynamics of Dexmedetomidine Administered as an Adjunct to Bupivacaine for Transversus Abdominis Plane Block in Patients Undergoing Lower Abdominal Cancer Surgery. J Pain Res. 2022 Jan 4;15:1-12. doi: 10.2147/JPR.S335806. eCollection 2022. PMID 35035233